CLINICAL TRIAL: NCT00743379
Title: A Phase 1/2, Multicenter, Dose-Escalation Study to Determine the Safety, Efficacy and Pharmacokinetics of TH-302 in Combination With A) Gemcitabine or B) Docetaxel or C) Pemetrexed in Patients With Advanced Solid Tumors
Brief Title: Dose-Escalation Study of TH-302 in Combination With A) Gemcitabine or B) Docetaxel or C) Pemetrexed to Treat Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Threshold Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-402
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Non-Small Cell Lung Cancer; Prostate Cancer; Pancreatic Cancer
Keywords: Phase 1/2; Advanced Solid Tumors; Hypoxia; Prodrug; Dose-Escalation; Evofosfamide
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms; Pancreatic Neoplasms; Hypoxia | interventions — TH 302

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): TH-302 in combination with Gemcitabine. 1,000 mg/m2 of Gemcitabine is administered IV over 30 minutes on Days 1, 8 and 15 of a 28-day cycle.
  Interventions: Drug: TH-302
- B (Experimental): TH-302 in combination with Docetaxel. 75 mg/m2 of Docetaxel is administered IV over 60 minutes on Day 1 of a 21-day cycle.
  Interventions: Drug: TH-302
- C (Experimental): TH-302 in combination with Pemetrexed. 500 mg/m2 of Pemetrexed is administered IV over 10 minutes on Day 1 of a 21-day cycle.
  Interventions: Drug: TH-302

INTERVENTIONS:
Drug: TH-302 — TH-302 will be administered by IV infusion over 30 minutes on Days 1, 8 and 15 of a 28- day cycle for Arm A and on Days 1 and 8 of a 21 day cycle for Arms B and C.

SUMMARY:
The purpose of this study is to determine if TH-302, in combination with A) Gemcitabine, or B) Docetaxel or C) Pemetrexed methotrexate, are safe and effective in the treatment of Pancreatic Cancer, Castrate-resistant Prostate Cancer, and Non-small Cell Lung Cancer, respectively.

DETAILED DESCRIPTION:
A broad range of tumors have been shown to contain significant numbers of hypoxic cells and hypoxia has been shown to be associated with a poor prognosis and an increase in resistance to chemotherapy and radiotherapy (Brizel 1997, Vaupel 2007, Shannon 2003).

It is likely that an agent that could effectively target hypoxic regions in tumors would improve efficacy when combined with standard chemotherapy or radiotherapy. TH-302 is activated at lower oxygen concentrations than other bioreductive prodrugs (Duan 2008) and tirapazamine, a hypoxic cytotoxin that has been extensively studied in both preclinical and clinical studies. This should result in an improved therapeutic ratio (tumor vs normal tissue toxicity) as compared with other bioreductive agents. Because TH-302 is expected to be minimally toxic to aerobic cancer cells, optimal efficacy would be expected when TH-302 is combined with treatments that are most effective under aerobic conditions such as radiotherapy and cytotoxic chemotherapy. Preclinical data have shown at least additive efficacy when TH-302 is combined with either docetaxel or gemcitabine. In order to minimize the risk of additive toxicity, TH-302 is not being evaluated in combination with alkylating agents.

ELIGIBILITY:
Gemcitabine + TH-302 Inclusion Criteria:

1. At least 18 years of age
2. Ability to understand the purposes and risks of the study and has signed a written informed consent form
3. Dose escalation subjects:

   a. Histologically or cytologically confirmed solid malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective OR solid malignancy for which monotherapy with gemcitabine is considered standard therapy b. Tumor progression after most recent therapy

   Dose expansion subjects:

   a. Locally advanced unresectable or metastatic pancreatic ductal adenocarcinoma proven either by histology (surgical biopsy) or cytology (CT- or endoscopic-guided) previously untreated with chemotherapy other than radiosensitizing doses of 5-fluorouracil
4. Recovered from toxicities of prior therapy to grade 0 or 1
5. Evaluable disease by RECIST criteria (at least one target or non-target lesion)
6. ECOG 0 or 1
7. Life expectancy of at least 3 months
8. Acceptable liver function:

   a. Bilirubin ≤ 1.5 times upper limit of normal b. AST (SGOT) and ALT (SGPT) ≤ 2.5xULN; if liver metastases are present, then ≤ 5xULN is allowed
9. Acceptable renal function:

   a. Serum creatinine ≤ ULN
10. Acceptable hematologic status:

    1. ANC ≥ 1500 cells/μL
    2. Platelet count ≥ 100,000/μL
    3. Hemoglobin ≥ 9.0 g/dL
11. All women of childbearing potential must have a negative serum pregnancy test and women and men subjects must agree to use effective means of contraception with their partner from entry into the study through 6 months after the last dose

Docetaxel + TH-302 Inclusion Criteria:

All Subjects:

1. At least 18 years of age
2. Ability to understand the purposes and risks of the study and has signed a written informed consent form
3. Dose escalation subjects ONLY:

   a. Histologically or cytologically confirmed solid malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective OR solid malignancy for which monotherapy with docetaxel would be appropriate b. Tumor progression after most recent therapy
4. Recovered from toxicities of prior therapy to grade 0 or 1
5. Evaluable disease by RECIST criteria (at least one target or non-target lesion) or evidence of disease progression for subjects with metastatic castrate-resistant prostate cancer
6. ECOG 0 or 1
7. Life expectancy of at least 3 months
8. Acceptable liver function:

   a. Bilirubin ≤ upper limit of normal b. AST (SGOT) and ALT (SGPT) ≤ 1.5x ULN with alkaline phosphatase ≤ 2.5x ULN
9. Acceptable renal function:

   a. Serum creatinine ≤ ULN
10. Acceptable hematologic status:

    1. ANC ≥ 1500 cells/μL
    2. Platelet count ≥ 100,000/μL
    3. Hemoglobin ≥ 9.0 g/dL
11. All women of childbearing potential must have a negative serum pregnancy test and women and men subjects must agree to use effective means of contraception with their partner from entry into the study through 6 months after the last dose

Expanded Cohort Subjects or dose-escalation subjects with metastatic castrate-resistant prostate cancer previously untreated with chemotherapy:

1. Histologically or cytologically confirmed adenocarcinoma of the prostate with clinical or radiologic evidence of metastatic disease
2. Disease progression during hormone therapy and received primary androgenablation therapy as maintenance
3. For subjects who have not had orchiectomy: serum testosterone concentration <50 ng/mL (<1.7 nmol/L); GnRH analog therapy must be continued during this study
4. If there has been antiandrogen withdrawal, it must have occurred at least 4 weeks before study enrollment (6 weeks for bicalutamide) OR in subjects who have had an antiandrogen added as second-line therapy and there was no response to the most recent antiandrogen therapy or if the PSA decline lasted ≤3 months, antiandrogen therapy must be discontinued for at least 2 weeks
5. Evidence of disease progression, manifested by at least one of the following:

   1. Rising PSA on at least 3 measurements at least 1 week apart
   2. Disease progression on physical examination or imaging studies (if progression is based on bone scan alone, there must be at least 2 new bone lesions)
6. Previously untreated with systemic chemotherapy
7. PSA at least 2 ng/mL

Expanded Cohort Subjects or dose-escalation subjects with second-line NSCLC:

1. Histological or cytological confirmation of NSCLC with stage IIIB or IV disease not amenable to curative therapy 2. Prior treatment with only one systemic chemotherapy regimen for advanced disease 3. Tumor progression after most recent therapy

Pemetrexed + TH-302 Inclusion Criteria:

All Subjects:

1. At least 18 years of age
2. Ability to understand the purposes and risks of the study and has signed a written informed consent form
3. Dose escalation subjects:

   a. Histologically or cytologically confirmed solid malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective OR solid malignancy for which monotherapy with pemetrexed is considered standard therapy b. Tumor progression after most recent therapy
4. Recovered from toxicities of prior therapy
5. Evaluable disease by RECIST criteria (at least one target or non-target lesion)
6. ECOG performance status of 0 or 1
7. Life expectancy of at least 3 months
8. Acceptable liver function:

   1. Bilirubin ≤ 1.5x ULN
   2. AST (SGOT) and ALT (SGPT) ≤ 2.5x ULN; if liver metastases are present, then ≤ 5x ULN is allowed
9. Acceptable renal function:

   a. Serum creatinine ≤ ULN and calculated CrCl ≥ 45 mL/min
10. Acceptable hematologic status:

    a. ANC ≥ 1500 cells/μL b. Platelet count ≥ 100,000/μL c. Hemoglobin ≥ 9.0 g/dL
11. All women of childbearing potential must have a negative serum pregnancy test and women and men subjects must agree to use effective means of contraception with their partner from entry into the study through 6 months after the last dose Expanded cohort subjects ONLY: Second-line NSCLC

1. Histological or cytological confirmation of NSCLC with stage IIIB or IV disease not amenable to curative therapy 2. Prior treatment with only one systemic chemotherapy regimen for advanced disease 3. Tumor progression after most recent therapy

Gemcitabine + TH-302 Exclusion Criteria:

All Subjects:

1. Prior treatment with more than 3 myelosuppressive cytotoxic chemotherapy regimens
2. Prior treatment with gemcitabine
3. Prior radiotherapy to more than 25% of the bone marrow
4. New York Heart Association (NYHA) Class III or IV, cardiac disease, myocardial infarction within 6 months prior to Day 1, unstable arrhythmia or symptomatic peripheral arterial vascular disease
5. Seizure disorders requiring anticonvulsant therapy
6. Symptomatic brain, leptomeningeal or epidural metastases, (unless previously treated and well controlled for a period of ≥ 3 months)
7. Previously treated malignancies, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancer from which the subject has been disease-free for at least 5 years
8. Severe chronic obstructive or other pulmonary disease with hypoxemia (requires supplementary oxygen, symptoms due to hypoxemia or oxygen saturation <90% by pulse oximetry after a 2 minute walk) or in the opinion of the investigator any physiological state likely to cause systemic or regional hypoxemia
9. Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery
10. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
11. Treatment with radiation therapy, surgery, chemotherapy, targeted therapies or hormones within 4 weeks prior to study entry
12. Prior therapy with an hypoxic cytotoxin
13. Subjects who participated in an investigational drug or device study within 28 days prior to study entry
14. Known infection with HIV, hepatitis B or C
15. Subjects who have exhibited allergic reactions to a structural compound, biological agent, or formulation (containing solutol and/or propylene glycol) similar to TH-302
16. Females who are pregnant or breast-feeding
17. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
18. Unwillingness or inability to comply with the study protocol for any reason Expanded cohort subjects ONLY: First-line advanced adenocarcinoma of the pancreas

1. Prior chemotherapy therapy for advanced disease other than radiosensitizing doses of 5-fluorouracil

Docetaxel + Prednisone + TH-302 Exclusion Criteria:

All Subjects:

1. Prior treatment with more than 3 myelosuppressive cytotoxic chemotherapy regimens
2. Prior treatment with docetaxel
3. Prior radiotherapy to more than 25% of the bone marrow unless radiotherapy was completed >5 years ago and there is not hematologic evidence of persistent bone marrow suppression
4. Uncontrolled pleural effusion or ascites
5. History of sensitivity to drugs formulated with polysorbate 80
6. New York Heart Association (NYHA) Class III or IV, cardiac disease, myocardial infarction within 6 months prior to Day 1, unstable arrhythmia or symptomatic peripheral arterial vascular disease
7. Seizure disorders requiring anticonvulsant therapy
8. Symptomatic brain, leptomeningeal or epidural metastases (unless previously treated and well controlled for a period of ≥ 3 months)
9. Ongoing CTCAE grade 2 or greater peripheral neuropathy
10. Previously treated malignancies, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancer from which the subject has been disease-free for at least 5 years
11. Severe chronic obstructive or other pulmonary disease with hypoxemia (requires supplementary oxygen, symptoms due to hypoxemia or oxygen saturation <90% by pulse oximetry after a 2 minute walk) or in the opinion of the investigator any physiological state likely to cause systemic or regional hypoxemia
12. Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery
13. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
14. Treatment with radiation therapy, surgery, chemotherapy, targeted therapies or hormones within 4 weeks prior to study entry
15. Prior therapy with an hypoxic cytotoxin
16. Subjects who participated in an investigational drug or device study within 28 days prior to study entry
17. Known active infection with HIV, hepatitis B or C
18. Subjects who have exhibited allergic reactions to a structural compound, biological agent, or formulation (containing solutol and/or propylene glycol) similar to TH-302
19. Females who are pregnant or breast-feeding
20. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
21. Unwillingness or inability to comply with the study protocol for any reason Expanded Cohort Subjects ONLY: Castrate-resistant prostate cancer

1. Prior treatment with cytotoxic chemotherapy or radioisotope therapy Expanded Cohort Subjects ONLY: Second-line NSCLC

1. More than one prior cytotoxic chemotherapy regimen for advanced disease
2. Weight loss of >10% body weight in the previous 6 weeks

Pemetrexed + TH-302 Exclusion Criteria:

All Subjects:

1. Prior treatment with more than 3 myelosuppressive cytotoxic chemotherapy regimens
2. Prior treatment with pemetrexed
3. Prior radiotherapy to more than 25% of the bone marrow
4. Inability to discontinue non-steroidal anti-inflammatory drugs for 5 days (long half-life) or 2 days (short half-life, if subject has CrCl <80 mL/min) before until 2 days following pemetrexed dosing
5. New York Heart Association (NYHA) Class III or IV, cardiac disease, myocardial infarction within 6 months prior to Day 1, unstable arrhythmia or symptomatic peripheral arterial vascular disease
6. Seizure disorders requiring anticonvulsant therapy
7. Symptomatic brain, leptomeningeal or epidural metastases (unless previously treated and well controlled for a period of ≥ 3 months)
8. Previously treated malignancies, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancer from which the subject has been disease-free for at least 5 years
9. Severe chronic obstructive or other pulmonary disease with hypoxemia (requires supplementary oxygen, symptoms due to hypoxemia or oxygen saturation <90% by pulse oximetry after a 2 minute walk) or in the opinion of the investigator any physiological state likely to cause systemic or regional hypoxemia
10. Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery
11. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
12. Treatment with radiation therapy, surgery, chemotherapy, targeted therapies or hormones within 4 weeks prior to study entry
13. Prior therapy with an hypoxic cytotoxin
14. Subjects who participated in an investigational drug or device study within 28 days prior to study entry
15. Known active infection with HIV, hepatitis B, or hepatitis C
16. Subjects who have exhibited allergic reactions to a structural compound, biological agent, or formulation (containing solutol and/or propylene glycol) similar to TH-302
17. Females who are pregnant or breast-feeding
18. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
19. Unwillingness or inability to comply with the study protocol for any reason Expanded Cohort Subjects ONLY: Second-line NSCLC

1. More than one prior cytotoxic chemotherapy regimen for advanced disease 2. Weight loss of >10% body weight in the previous 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-08; Primary Completion 2013-07 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To determine the MTD and DLT(s) of TH-302 when used in combination with A) Gemcitabine or B) Docetaxel or C) Pemetrexed in patients with advanced solid tumors | Two years

SECONDARY OUTCOMES:
To establish the pharmacokinetics of TH-302 , gemcitabine, pemetrexed and docetaxel when used in each of the combinations assessed | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Infante, MD, Principal Investigator — SCRI Development Innovations, LLC; Mitesh Borad, MD, Principal Investigator — Mayo Clinic
Locations (11):
- United States (11):
  - Mayo Clinic Cancer Center, Scottsdale, Arizona
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - Indiana University Cancer Center, Indianapolis, Indiana
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - UT Health Science Center, San Antonio, Texas
  - Northwest Medical Specialties, Tacoma, Washington
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Result] Borad MJ, Reddy SG, Bahary N, Uronis HE, Sigal D, Cohn AL, Schelman WR, Stephenson J Jr, Chiorean EG, Rosen PJ, Ulrich B, Dragovich T, Del Prete SA, Rarick M, Eng C, Kroll S, Ryan DP. Randomized Phase II Trial of Gemcitabine Plus TH-302 Versus Gemcitabine in Patients With Advanced Pancreatic Cancer. J Clin Oncol. 2015 May 1;33(13):1475-81. doi: 10.1200/JCO.2014.55.7504. Epub 2014 Dec 15. PMID 25512461
- See also: Threshold Pharmaceuticals Company Website — http://www.thresholdpharm.com